CLINICAL TRIAL: NCT06489613
Title: Screening for Monoclonal Gammopathy in Individuals Undergoing Physical Examinations Using iMS-LC Assay Technology.
Status: Not yet recruiting | Type: Observational
Sponsor: Jian Li (Other)
Responsible Party: Sponsor-Investigator, Jian Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: iMS-LC Assay
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: M Protein; Monoclonal Gammopathy; Monoclonal Gammopathy of Undetermined Significance
Keywords: M protein; Monoclonal gammopathy of unknown significance
MeSH Terms: conditions — Paraproteinemias; Monoclonal Gammopathy of Undetermined Significance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Clinical residual serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical patients: Residual plasma specimens for iMS-LC Assay to detect M protein
  Interventions: Diagnostic Test: M protein detection by iMS-LC Assay
- Individuals undergoing routine physical examinations: Residual plasma specimens for iMS-LC Assay to detect M protein
  Interventions: Diagnostic Test: M protein detection by iMS-LC Assay

INTERVENTIONS:
Diagnostic Test: M protein detection by iMS-LC Assay — iMS-LC Assay (intact M-protein Screening-Light Chain Assay) technology is a new method for the specific identification of M-proteins in peripheral blood, based on mass spectrometry recognition of intact clonal immunoglobulin light chains. Combined with AI algorithm models, M-proteins can be easily distinguished from the polyclonal background, enabling automated identification and quantitative analysis of M-proteins.
  Previous studies have shown that the detection limit of the iMS-LC Assay is several times higher than that of IFE. Additionally, the iMS-LC Assay requires only 5 μL of peripheral blood serum for detection, offering advantages over traditional methods in terms of higher sensitivity, non-invasiveness, lower sample volume requirements, reduced detection costs, and higher throughput.

SUMMARY:
iMS-LC Assay (intact M-protein Screening-Light Chain Assay) is a new technology based on mass spectrometry identification of intact clonal immunoglobulin light chains for the specific detection of M-proteins in peripheral blood.

The investigators propose to conduct a prospective, single-center observational study to screen for M-proteins in the peripheral blood of individuals undergoing routine physical examinations using iMS-LC Assay technology. The goals of this observational study are : (1) to evaluate the diagnostic efficacy of detecting peripheral blood M-proteins using the iMS-LC Assay method; and (2) to determine the prevalence of MGUS in the population undergoing routine physical examinations based on mass spectrometry screening.

Initially, the investigators will collect clinical patient samples continuously and conduct a diagnostic trial of the iMS-LC Assay, using the clinical methods SPEP + SIFE + FLC as the gold standard. Based on the diagnostic performance of the iMS-LC Assay, the investigators will then screen for M-proteins in continuous samples from individuals undergoing routine physical examinations, to further determine the prevalence of MGUS in this population based on mass spectrometry screening.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical patients:

   * ≥18 years old;
   * have concurrent SPEP + SIFE + FLC test results.
2. Individuals undergoing routine physical examinations:

   * ≥30 years old;
   * have concurrent SPEP test results.

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Clinical patients: 600 continuous outpatients/inpatients diagnosed with or suspected of having monoclonal gammopathy.
  2. 15,000 continuous individuals undergoing routine physical examinations.
Sampling Method: Non-Probability Sample
Enrollment: 15600 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy of the iMS-LC Assay | 2024-07 to 2024-10
  Using any positive result from SPEP + SIFE + FLC as the gold standard, we will obtain the diagnostic performance parameters of the iMS-LC Assay for M-protein detection, including sensitivity, specificity, kappa value, likelihood ratio, and predictive values.
Prevalence of MGUS in the population undergoing routine physical examinations | 2024-07 to 2024-12
  The prevalence of MGUS in the population undergoing routine physical examinations based on mass spectrometry screening.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Murray DL, Puig N, Kristinsson S, Usmani SZ, Dispenzieri A, Bianchi G, Kumar S, Chng WJ, Hajek R, Paiva B, Waage A, Rajkumar SV, Durie B. Mass spectrometry for the evaluation of monoclonal proteins in multiple myeloma and related disorders: an International Myeloma Working Group Mass Spectrometry Committee Report. Blood Cancer J. 2021 Feb 1;11(2):24. doi: 10.1038/s41408-021-00408-4. PMID 33563895
- [Background] Kohlhagen M, Dasari S, Willrich M, Hetrick M, Netzel B, Dispenzieri A, Murray DL. Automation and validation of a MALDI-TOF MS (Mass-Fix) replacement of immunofixation electrophoresis in the clinical lab. Clin Chem Lab Med. 2020 Aug 3;59(1):155-163. doi: 10.1515/cclm-2020-0581. PMID 32745067
- [Background] Dasari S, Kohlhagen MC, Dispenzieri A, Willrich MAV, Snyder MR, Kourelis TV, Lust JA, Mills JR, Kyle RA, Murray DL. Detection of Plasma Cell Disorders by Mass Spectrometry: A Comprehensive Review of 19,523 Cases. Mayo Clin Proc. 2022 Feb;97(2):294-307. doi: 10.1016/j.mayocp.2021.07.024. Epub 2021 Dec 7. PMID 34887112
- [Background] Keren DF, Bocsi G, Billman BL, Etzell J, Faix JD, Kumar S, Lipe B, McCudden C, Montgomery R, Murray DL, Rai AJ, Redondo TC, Souter L, Ventura CB, Ansari MQ. Laboratory Detection and Initial Diagnosis of Monoclonal Gammopathies. Arch Pathol Lab Med. 2022 May 1;146(5):575-590. doi: 10.5858/arpa.2020-0794-CP. PMID 34347866